CLINICAL TRIAL: NCT04583423
Title: A Phase 2b Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of MK-3655 in Individuals With Pre-cirrhotic Nonalcoholic Steatohepatitis.
Brief Title: A Study of MK-3655 in Individuals With Pre-cirrhotic Nonalcoholic Steatohepatitis (NASH) (MK-3655-001)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Business reasons
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3655-001; MK-3655-001 (Other: Merck Protocol Number); jRCT2051200083 (Registry Identifier: jRCT); 2019-003048-63 (EudraCT Number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Results first posted 2024-04-29 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Nonalcoholic Steatohepatitis
Keywords: Non-alcoholic fatty liver disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- MK-3655 50 mg (Experimental): Following a 2-week placebo run-in, participants will receive MK-3655 50 mg by subcutaneous (SC) injection once every 4 weeks (Q4W) for 52 weeks.
  Interventions: Drug: MK-3655
- MK-3655 100 mg (Experimental): Following a 2-week placebo run-in, participants will receive MK-3655 100 mg by SC injection Q4W for 52 weeks.
  Interventions: Drug: MK-3655
- MK-3655 300 mg (Experimental): Following a 2-week placebo run-in, participants will receive MK-3655 300 mg by SC injection Q4W for 52 weeks.
  Interventions: Drug: MK-3655
- Placebo (Placebo Comparator): Following a 2-week placebo run-in, participants will receive Placebo by SC injection Q4W for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-3655 — MK-3655 50, 100 or 300 dose for injection
  Other Names: NGM313
  Arms: MK-3655 100 mg; MK-3655 300 mg; MK-3655 50 mg
Drug: Placebo — Matching placebo to MK-3655
  Arms: Placebo

SUMMARY:
This study will evaluate the effect of each dose of MK-3655 versus placebo on the percentage of individuals with NASH resolution without worsening of fibrosis after 52 weeks. The primary hypothesis of the study is that at least 1 dose of MK-3655 is superior to placebo with respect to the percentage of individuals with NASH resolution without worsening of fibrosis after 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Has histological confirmation of NASH
* Is a male or female aged 18 years to 80 years (in Japan and Taiwan aged 20 to 80 years)
* Has a body mass index (BMI) ≥25 kg/m^2 and ≤50 kg/m^2 and stable weight for the past 3 months
* Has no history of Type 2 diabetes mellitus (T2DM) OR a history of T2DM controlled by diet or stable doses of antihyperglycemic agents (AHAs)
* Contraceptive use by male participants should be consistent with local regulations.
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and she is not a woman of child-bearing potential (WOCBP) OR she is a WOCBP and uses a contraceptive method that is highly effective during the intervention period and for at least 16 weeks after the last dose of study intervention.

Exclusion Criteria

* Has presence of cirrhosis on liver biopsy
* Has Type 1 diabetes
* Has a history of malignancy, unless cancer free ≥5 years, or is under evaluation for active or suspected malignancy except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer
* Has a history of bariatric surgery ≤5 years before study participation
* Has undergone a major surgical procedure ≤3 months before study participation or has major surgery planned during the study
* Has a history or evidence of chronic liver disease other than NASH. Individuals with a history of Hepatitis B or C may be eligible for participation.
* Has significant systemic or major illnesses other than liver disease, including recent events (≤6 months before study entry) of congestive heart failure, unstable coronary artery disease, arterial revascularization, pulmonary disease, renal failure, stroke, transient ischemic attack, or organ transplantation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Actual)
Dates: Start 2020-11-11 (Actual); Primary Completion 2023-04-13 (Actual); Study Completion 2023-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Merck Sharp & Dohme LLC
Locations (180):
- United States (48):
  - Adobe Clinical Research, LLC ( Site 2644), Tucson, Arizona
  - Arizona Liver Health ( Site 9026), Tucson, Arizona
  - Del Sol Research Management ( Site 2674), Tucson, Arizona
  - Arkansas Gastroenterology - North Little Rock ( Site 9015), North Little Rock, Arkansas
  - Hope Clinical Research, Inc. ( Site 2601), Canoga Park, California
  - Velocity Clinical Research, Huntington Park ( Site 9022), Huntington Park, California
  - UCSD - Altman Clinical and Translational Research Institute -UC San Diego NAFLD Research Center ( Si, La Jolla, California
  - Ruane Clinical Research Group, Inc ( Site 9014), Los Angeles, California
  - Velocity Clinical Research, Westlake ( Site 9013), Los Angeles, California
  - Catalina Research Institute, LLC ( Site 2643), Montclair, California
  - Velocity Clinical Research, Panorama City ( Site 9001), Panorama City, California
  - California Liver Research Institute ( Site 9025), Pasadena, California
  - Quest Clinical Research ( Site 9011), San Francisco, California
  - Velocity Clinical Research, Santa Ana ( Site 9002), Santa Ana, California
  - Peak Gastroenterology Associates ( Site 2645), Colorado Springs, Colorado
  - Top Medical Research, Inc ( Site 2673), Cutler Bay, Florida
  - Covenant Metabolic Specialists, LLC ( Site 9027), Fort Myers, Florida
  - North Florida South Georgia Veterans Health System ( Site 2613), Gainesville, Florida
  - Indago Research and Health Center Inc ( Site 2610), Hialeah, Florida
  - Sweet Hope Research Specialty Inc ( Site 2660), Hialeah, Florida
  - Genoma Research Group, Inc. ( Site 2669), Miami, Florida
  - Floridian Clinical Research, LLC ( Site 2656), Miami Lakes, Florida
  - Ocean Blue Medical Research Center Inc ( Site 2667), Miami Springs, Florida
  - Sensible Healthcare Llc ( Site 2607), Ocoee, Florida
  - Synexus Research ( Site 2672), Orlando, Florida
  - Southeast Clinical Research Center ( Site 9003), Dalton, Georgia
  - The University of Iowa ( Site 2655), Iowa City, Iowa
  - Legacy Clinical Solutions: Tandem Clinical Research, LLC ( Site 2650), Marrero, Louisiana
  - The National Diabetes & Obesity Research Institute ( Site 9017), Biloxi, Mississippi
  - Kansas City Research Institute ( Site 9018), Kansas City, Missouri
  - Excel Clinical Research, LLC ( Site 2603), Las Vegas, Nevada
  - Velocity Clinical Research, Syracuse ( Site 9016), East Syracuse, New York
  - NYU Langone Health, New York ( Site 2627), New York, New York
  - Hillmont G.I. ( Site 9019), Flourtown, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, LTD ( Site 9020), Lancaster, Pennsylvania
  - Regional Gastroenterology Associates of Lancaster, LTD ( Site 9004), Wyomissing, Pennsylvania
  - Premier Medical Group ( Site 9010), Clarksville, Tennessee
  - Texas Clinical Research Institute ( Site 2619), Arlington, Texas
  - The Liver Institute at Methodist Dallas Medical Center ( Site 2638), Dallas, Texas
  - DHR Health Institute for Research and Development ( Site 9006), Edinburg, Texas
  - South Texas Research Institute ( Site 9012), Edinburg, Texas
  - Baylor College of Medicine - Advanced Liver Therapies ( Site 2670), Houston, Texas
  - The Crofoot Research Center, Inc. ( Site 2611), Houston, Texas
  - Quality Research ( Site 9024), San Antonio, Texas
  - American Research Corporation at Texas Liver Institute ( Site 2634), San Antonio, Texas
  - Clinical Trials of Texas, LLC ( Site 2614), San Antonio, Texas
  - Impact Research Institute ( Site 2685), Waco, Texas
  - Virginia Commonwealth University Health System ( Site 2657), Richmond, Virginia
- Argentina (9):
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0010), Mar del Plata, Buenos Aires
  - Hospital Universitario Austral ( Site 0003), Pilar, Buenos Aires
  - DIM Clínica Privada ( Site 0011), Ramos Mejía, Buenos Aires
  - Hospital Británico de Buenos Aires ( Site 0002), Buenos Aires, Buenos Aires F.D.
  - Glenny Corp. S.A.-CLINICAL RESEARCH ( Site 0013), Buenos Aires, Buenos Aires F.D.
  - Hospital Italiano de Buenos Aires-Hepatology ( Site 0014), Ciudad de Buenos Aires, Buenos Aires F.D.
  - Hospital Provincial del Centenario ( Site 0007), Rosario, Santa Fe Province
  - Hospital Aleman ( Site 0009), Buenos Aires
  - Clinica de nefrologia urologia y enfermedades cardiovasculares ( Site 0008), Santa Fe
- Australia (3):
  - Royal Prince Alfred Hospital ( Site 0102), Camperdown, New South Wales
  - St George Hospital ( Site 0104), Kogarah, New South Wales
  - Flinders Medical Centre ( Site 0107), Bedford Park, South Australia
- Canada (3):
  - GIRI GI Research Institute - Vancouver ( Site 0404), Vancouver, British Columbia
  - University Health Network - Toronto General Hospital ( Site 0401), Toronto, Ontario
  - McGill University Health Centre ( Site 0400), Montreal, Quebec
- Chile (6):
  - Hospital San Juan de Dios de La Serena ( Site 0500), La Serena, Coquimbo Region
  - Clinical Research Chile SpA ( Site 0506), Valdivia, Los Ríos Region
  - Enroll SpA ( Site 0508), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 0501), Santiago, Region M. de Santiago
  - Centro de Investigaciones Clinicas Vina del Mar ( Site 0502), Viña del Mar, Región de Valparaíso
  - Hospital Regional de Concepcion ( Site 0505), Concepción, Región del Biobío
- China (6):
  - Beijing YouAn Hospital, Capital Medical University ( Site 0605), Beijing, Beijing Municipality
  - Chongqing Three Gorges Central Hospital ( Site 0618), Wanzhou District, Chongqing Municipality
  - The First People's Hospital of Foshan-Infection Department ( Site 0612), Foshan, Guangdong
  - General Hospital of Ningxia Medical University ( Site 0607), Yinchuan, Ningxia
  - Xinhua Hospital Affiliated to Jiaotong University School of Medicine ( Site 0602), Shanghai, Shanghai Municipality
  - The Affiliated Hospital of Hangzhou Normal University ( Site 0600), Hangzhou, Zhejiang
- Fundacion Santa Fe de Bogota ( Site 0705), Bogotá, Bogota D.C., Colombia
- France (13):
  - CHU de Nice Hopital de l Archet II ( Site 0800), Nice, Alpes-Maritimes
  - hopital haut leveque chu de bordeaux-Service d'Hépato-gastroentérologie ( Site 0805), Pessac, Aquitaine
  - Hopital de la Croix-Rousse ( Site 0809), Lyon, Auvergne
  - CHU Dijon Bourgogne - Hopital F. Mitterrand ( Site 0816), Dijon, Bourgogne-Franche-Comté
  - CHU Besançon ( Site 0806), Besançon, Franche-Comte
  - Centre Hospitalier et Universitaire Dupuytren ( Site 0810), Limoges, Haute-Vienne
  - Hôpital Beaujon ( Site 0804), Clichy, Hauts-de-Seine
  - C.H.U. Nancy Hopital de Brabois ( Site 0803), Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Hôpital Claude Huriez ( Site 0811), Lille, Nord
  - Hopital Henri Mondor ( Site 0808), Créteil, Val-de-Marne
  - A.P.H. Paris, Hopital Saint Antoine ( Site 0807), Paris
  - Hopital de la Pitie Salpetriere ( Site 0813), Paris
  - Hopitaux Universitaires Paris Centre-Hopital Cochin ( Site 0812), Paris
- Germany (5):
  - Universitaetsklinikum Freiburg ( Site 0446), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitätsklinikum Frankfurt-Medizinische Klinik 1 ( Site 0445), Frankfurt am Main, Hesse
  - Johannes Gutenberg Universitat Mainz ( Site 0442), Mainz, Rhineland-Palatinate
  - Universitaetsklinikum Leipzig ( Site 0447), Leipzig, Saxony
  - Charite Universitaetsmedizin Berlin ( Site 0443), Berlin
- Hippokration University Hopsital-4th Department of Internal Medicine ( Site 3300), Thessaloniki, Central Macedonia, Greece
- Hong Kong (3):
  - Queen Mary Hospital ( Site 1003), Hong Kong
  - Prince of Wales Hospital ( Site 1001), Shatin
  - Prince of Wales Hospital ( Site 1002), Shatin
- Israel (7):
  - Rambam Medical Center ( Site 1201), Haifa
  - Carmel Medical Center ( Site 1203), Haifa
  - Shaare Zedek Medical Center ( Site 1205), Jerusalem
  - Rabin Medical Center ( Site 1204), Petah Tikva
  - Chaim Sheba Medical Center ( Site 1200), Ramat Gan
  - Maccabi Health Services - Ramat Hasharon ( Site 1206), Ramat HaSharon
  - Sourasky Medical Center ( Site 1202), Tel Aviv
- Italy (4):
  - IRCCS Istituto Clinico Humanitas di Rozzano ( Site 1303), Rozzano, Lombardy
  - A O U Policlinico di Modena ( Site 1307), Modena
  - Azienda Ospedaliera Policlinico Umberto I ( Site 1300), Roma
  - Azienda Ospedaliera Universitaria Integrata Verona ( Site 1301), Verona
- Japan (19):
  - Aichi Medical University Hospital ( Site 1402), Nagakute, Aichi-ken
  - Ehime University Hospital ( Site 1417), Tōon, Ehime
  - Ogaki Municipal Hospital ( Site 1409), Ōgaki, Gifu
  - Hokkaido P.W.F.A.C Sapporo-Kosei General Hospital ( Site 1404), Sapporo, Hokkaido
  - Kanazawa University Hospital ( Site 1419), Kanazawa, Ishikawa-ken
  - Kagawa University Hospital ( Site 1414), Kita-gun, Kagawa-ken
  - Kagawa Prefectural Central Hospital-liver intemal medicine ( Site 1416), Takamatsu, Kagawa-ken
  - Shinyurigaoka General Hospital ( Site 1420), Kawasaki, Kanagawa
  - Yokohama City University Hospital ( Site 1411), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 1407), Kashihara, Nara
  - Saiseikai Suita Hospital ( Site 1403), Suita, Osaka
  - Fukui-ken Saiseikai Hospital ( Site 1410), Fukui
  - Gifu Municipal Hospital ( Site 1408), Gifu
  - Hiroshima University Hospital ( Site 1413), Hiroshima
  - Kagoshima University Hospital ( Site 1418), Kagoshima
  - University Hospital, Kyoto Prefectural University of Medicine ( Site 1405), Kyoto
  - Kawasaki Medical School General Medical Center ( Site 1412), Okayama
  - Osaka Metropolitan University Hospital ( Site 1415), Osaka
  - Toranomon Hospital ( Site 1401), Tokyo
- Hospital Kuala Lumpur-Gastroenterology Department ( Site 2701), Kuala Lumpur, Malaysia
- Mexico (5):
  - Centro de Investigacion Medico Biologica y Terapia Avanzada SC ( Site 1511), Guadalajara, Jalisco
  - Centro de Investigacion Medica de Occidente S.C. ( Site 1514), Zapopan, Jalisco
  - Medica Sur-Clinica de Enfermedades Digestivas y Obesidad ( Site 1515), Mexico City, Mexico City
  - Medical Care and Research S.A. de C.V. ( Site 1506), Mérida, Yucatán
  - Centro de Investigacion y Gastroenterologia SC ( Site 1503), Mexico City
- New Zealand (3):
  - Christchurch Hospital ( Site 1602), Christchurch, Canterbury
  - Auckland Clinical Studies Limited ( Site 1600), Auckland
  - Middlemore Clinical Trials ( Site 1601), Auckland
- Puerto Rico (3):
  - Pan American Center for Oncology Trials ( Site 3102), Rio Piedras
  - Klinical Investigations Group ( Site 3100), San Juan
  - FDI Clinical Research ( Site 3101), San Juan
- Russia (9):
  - City Clinical Hospital named V.M.Buyanova ( Site 1922), Moscow, Moscow
  - Russian University of People Friendship ( Site 1907), Moscow, Moscow
  - Nephrology Clinic of Internal and Prof. Diseases n.a.E.M.Tareev ( Site 1906), Moscow, Moscow
  - Center targetnoy therapy-Gastroenterology ( Site 1918), Moscow, Moscow
  - Medical Rehabilitation Center ( Site 1904), Moscow, Moscow
  - SPb State Budgetary Institution Health Care City Policlinic 17 ( Site 1910), Saint Petersburg, Sankt-Peterburg
  - Scientific research center ECO-security ( Site 1920), Saint Petersburg, Sankt-Peterburg
  - Surgical Clinic "Parada" ( Site 1921), Saint Petersburg, Sankt-Peterburg
  - LLC Astarta ( Site 1912), Saint Petersburg, Sankt-Peterburg
- South Korea (9):
  - Seoul National University Bundang Hospital-Internal Medicine ( Site 2005), Seongnam, Kyonggi-do
  - Pusan National University Hospital-Internal Medicine ( Site 2010), Busan, Pusan-Kwangyokshi
  - Chungang University Hospital ( Site 2007), Dongjak-gu, Seoul
  - Asan Medical Center ( Site 2001), Songpagu, Seoul
  - Inha University Hospital-Gastroenterolgy/Hepatology ( Site 2006), Incheon
  - Seoul National University Hospital ( Site 2003), Seoul
  - Hanyang University Seoul Hospital ( Site 2002), Seoul
  - Samsung Medical Center-Gastroenterology/Internal Medicine ( Site 2008), Seoul
  - Korea University Guro Hospital ( Site 2004), Seoul
- Spain (6):
  - Hospital Universitario Marqués de Valdecilla-Gastroenterology and Hepatology ( Site 2106), Santander, Cantabria
  - Hospital Clinico Universitario de Santiago ( Site 2104), Santiago de Compostela, La Coruna
  - Hospital Universitario Puerta de Hierro-Majadahonda ( Site 2100), Majadahonda, Madrid
  - Hospital Universitario Virgen del Rocio ( Site 2105), Seville, Sevilla
  - Hospital Universitari Vall d Hebron ( Site 2101), Barcelona
  - Hospital Clinic de Barcelona ( Site 2102), Barcelona
- Sweden (2):
  - Karolinska Universitetssjukhuset Huddinge ( Site 2900), Huddinge, Stockholm County
  - Akademiska sjukhuset ( Site 2901), Uppsala, Uppsala County
- Taiwan (7):
  - Chiayi Christian Hospital ( Site 2308), Chiayi City, Chiayi
  - Chung Shan Medical University Hospital ( Site 2307), Taichung, Taichung
  - Chang Gung Memorial Hospital - Linkou Branch ( Site 2305), Taoyuan, Taoyuan
  - Kaohsiung Medical University Chung-Ho Memorial Hospital ( Site 2302), Kaohsiung City
  - Taichung Veterans General Hospital ( Site 2306), Taichung
  - National Cheng Kung University Hospital ( Site 2304), Tainan
  - National Taiwan University Hospital ( Site 2301), Taipei
- Turkey (Türkiye) (7):
  - Hacettepe Uni. Ic Hastaliklari Anabilim Dali, Nefroloji BD ( Site 2403), Ankara
  - Gazi University Medical Faculty ( Site 2405), Ankara
  - Ankara University Cebeci Research and Application Hospital ( Site 2406), Ankara
  - Bezmialem Vakf Üniversitesi-Gastroenterology ( Site 2402), Istanbul
  - Istanbul Universitesi Tip Fakultesi Hastanesi ( Site 2401), Istanbul
  - Marmara Universitesi Pendik Egitim ve Arastirma Hastanesi ( Site 2400), Istanbul
  - Ege University Medical Faculty ( Site 2404), Izmir

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Raji A, Gantz I, Crutchlow M, Flynn H, Xu L, Rodgers AJ, Krishnan R, Rizk ML, Hu S, Kaufman KD, Engel SS; MK-3655 P001 Study Group. Clinical Trial: A Phase 2b Study to Evaluate the Efficacy and Safety of MK-3655 in Individuals With Pre-Cirrhotic MASH. Aliment Pharmacol Ther. 2025 Apr;61(7):1152-1162. doi: 10.1111/apt.70038. Epub 2025 Feb 21. PMID 39984821
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Males and females with pre-cirrhotic Nonalcoholic Steatohepatitis (NASH) aged 18 to 80 years (in Japan and Taiwan, aged 20 to 80 years were randomized in this study
Groups:
- MK-3655 50 mg: Following a 2-week placebo run-in, participants received MK-3655 50 mg by subcutaneous (SC) injection once every 4 weeks (Q4W) for 52 weeks.
- MK-3655 100 mg: Following a 2-week placebo run-in, participants received MK-3655 100 mg by SC injection Q4W for 52 weeks.
- MK-3655 300 mg: Following a 2-week placebo run-in, participants received MK-3655 300 mg by SC injection Q4W for 52 weeks.
- Placebo: Following a 2-week placebo run-in, participants received placebo by SC injection Q4W for 52 weeks.
Period: Overall Study
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Started | 45 | 48 | 46 | 44
Received 1st Dose | 45 | 47 | 46 | 44
Completed | 10 | 11 | 8 | 8
Not Completed | 35 | 37 | 38 | 36
Not completed — Lost to Follow-up | 0 | 1 | 0 | 2
Not completed — Study Terminated by Sponsor | 32 | 35 | 36 | 33
Not completed — Withdrawal by Subject | 3 | 1 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- MK-3655 50 mg: Following a 2-week placebo run-in, participants received MK-3655 50 mg by SC injection Q4W for 52 weeks.
- Total: Total of all reporting groups
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo | Total
Number analyzed (Participants) | 45 | 48 | 46 | 44 | 183
Age, Continuous [Mean (Standard Deviation); unit: Years] | 59.6 (8.9) | 54.3 (12.3) | 56.6 (11.3) | 55.8 (10.1) | 56.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 20 | 23 | 19 | 87
  Male | 20 | 28 | 23 | 25 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 13 | 17 | 18 | 60
  Not Hispanic or Latino | 33 | 34 | 28 | 25 | 120
  Unknown or Not Reported | 0 | 1 | 1 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 15 | 18 | 16 | 16 | 65
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1 | 0 | 2
  Black or African American | 3 | 2 | 1 | 1 | 7
  White | 26 | 28 | 27 | 26 | 107
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Baseline Fibrosis Stage [Count of Participants; unit: Participants] — The NASH Clinical Research Network (CRN) scoring system assesses NASH activity and fibrosis stage based on the following scoring scales: lobular inflammation score (0-3); hepatocyte ballooning score (0-2); steatosis score (0-3); and fibrosis score (0-4). The Nonalcoholic Fatty Liver Disease (NAFLD) Activity Score (NAS) was calculated as the unweighted sum of the scores for inflammation, ballooning, and steatosis and ranged from 0-8 (highest activity).
  Participants
    Stage 2 | 21 | 22 | 21 | 21 | 85
    Stage 3 | 24 | 26 | 25 | 23 | 98
Percent Liver Fat Content [Count of Participants; unit: Participants] — Assessed via Magnetic Resonance Imaging-Estimated Proton Density Fat Fraction (MRI-PDFF), a highly accurate noninvasive measure of the proportion of fat content of a tissue
  Participants
    <20% | 30 | 23 | 30 | 31 | 114
    ≥ 20% | 15 | 25 | 16 | 13 | 69
Type 2 Diabetes Mellitus (T2DM) [Count of Participants; unit: Participants]
  Yes | 22 | 25 | 25 | 24 | 96
  No | 23 | 23 | 21 | 20 | 87
Region [Count of Participants; unit: Participants]
  Japan | 11 | 12 | 11 | 11 | 45
  East Asia excluding Japan | 6 | 5 | 5 | 5 | 21
  Other | 28 | 31 | 30 | 28 | 117

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Nonalcoholic Steatohepatitis (NASH) Resolution Without Worsening of Fibrosis After 52 Weeks
Description: The NASH Clinical Research Network (CRN) scoring system evaluated by Blinded Independent Central Review (BICR) was used to assess treatment response. The NASH CRN scoring scales were: lobular inflammation score (0-3); hepatocyte ballooning score (0-2); steatosis score (0-3); and fibrosis score (0-4). NASH resolution was defined as a score of 0-1 for inflammation, 0 for ballooning, and any grade of steatosis.
Time Frame: Week 52
Population: Full Analysis Set (FAS) population, which consisted of all randomized participants who had at least 1 injection of study intervention and had at least 1 assessment
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Number analyzed (Participants) | 18 | 21 | 17 | 17
Percentage of Participants | 16.7 | 14.3 | 17.6 | 5.9
Statistical Analysis 1: Comparison: MK-3655 50 mg vs Placebo; Test type: Other; p = 0.3504, Miettinen and Nurminen's method; Stratified by concurrent diagnosis of T2DM at the time of randomization and fibrosis score and using Cochran-Mantel-Haenszel weighting scheme; Difference in Percentages = 10.4, 95% CI 2-sided [-13.4 to 35.1] — Difference=% 50-mg MK-3655 minus % placebo
Statistical Analysis 2: Comparison: MK-3655 100 mg vs Placebo; Test type: Other; p = 0.3730, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 9.2, 95% CI 2-sided [-15.6 to 32.1] — Difference=% 100-mg MK-3655 minus % placebo
Statistical Analysis 3: Comparison: MK-3655 300 mg vs Placebo; Test type: Other; p = 0.1428, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 15.4, 95% CI 2-sided [-8.5 to 42.3] — Difference=% 300-mg MK-3655 minus % placebo

2. Primary Outcome: Percentage of Participants Who Experienced an Adverse Event (AE)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it was considered related to the medical treatment or procedure, that occurred during the course of the study.
Time Frame: Up to 64 weeks
Population: All Participants as Treated (APaT) population, which included all randomized participants who received at least 1 injection of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 44
Percentage of Participants | 73.3 | 70.2 | 76.1 | 77.3

3. Primary Outcome: Percentage of Participants Discontinuing Study Medication Due to an AE
Description: as for outcome 2
Time Frame: Up to 52 weeks
Population: APaT population, which included all randomized participants who received at least 1 injection of study intervention
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Number analyzed (Participants) | 45 | 47 | 46 | 44
Percentage of Participants | 2.2 | 0 | 0 | 0

4. Secondary Outcome: Mean Percent Relative Reduction From Baseline in Liver Fat Content (LFC) After 24 Weeks
Description: LFC % was measured by Magnetic Resonance Imaging-Estimated Proton Density Fat Fraction (MRI-PDFF) and evaluated by BICR. MRI-PDFF is a highly accurate noninvasive measure of the proportion of fat content of a tissue.
Time Frame: Baseline and Week 24
Population: FAS population, which consisted of all randomized participants who had at least 1 injection of study intervention and had at least 1 assessment
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Number analyzed (Participants) | 33 | 36 | 37 | 31
Percent Change | 30.1 [17.5 to 42.7] | 30.0 [18.2 to 41.8] | 37.2 [25.5 to 48.8] | 11.0 [-0.9 to 23.0]
Statistical Analysis 1: Comparison: MK-3655 50 mg vs Placebo; Test type: Other; Difference in Least Square (LS) Means = 19.1, 95% CI 2-sided [1.7 to 36.4] — Difference=LS Mean 50 mg minus LS Mean Placebo
Statistical Analysis 2: Comparison: MK-3655 100 mg vs Placebo; Test type: Other; Difference in LS Means = 19.0, 95% CI 2-sided [2.2 to 35.8] — Difference=LS Mean 100 mg minus LS Mean Placebo
Statistical Analysis 3: Comparison: MK-3655 300 mg vs Placebo; Test type: Other; Difference in LS Means = 26.1, 95% CI 2-sided [9.5 to 42.8] — Difference=LS Mean 300 mg minus LS Mean Placebo

5. Secondary Outcome: Percentage of Participants With ≥1 Stage Improvement in Fibrosis Without Worsening of Steatohepatitis Assessed With the NASH CRN Scoring System After 52 Weeks
Description: Participants were evaluated with the NASH CRN scoring system with BICR with ≥1 stage improvement in fibrosis without worsening of steatohepatitis defined as no increase in the ballooning, inflammation, or steatosis scores.
Time Frame: Week 52
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Number analyzed (Participants) | 18 | 21 | 17 | 17
Percentage of Participants | 22.2 | 38.1 | 29.4 | 17.6
Statistical Analysis 1: Comparison: MK-3655 50 mg vs Placebo; Test type: Other; p = 0.8978, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 1.6, 95% CI 2-sided [-26.5 to 30.3] — Difference=% 50 mg minus % Placebo
Statistical Analysis 2: Comparison: MK-3655 100 mg vs Placebo; Test type: Other; p = 0.1869, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Parentages = 20.0, 95% CI 2-sided [-10.6 to 46.4] — Difference=% 100 mg minus % Placebo
Statistical Analysis 3: Comparison: MK-3655 300 mg vs Placebo; Test type: Other; p = 0.5636, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 8.5, 95% CI 2-sided [-22.1 to 38.5] — Difference=% 300 mg minus % Placebo

6. Secondary Outcome: Percentage of Participants With ≥2 Point Improvement in NAS With ≥1 Point Improvement in Inflammation or Ballooning Without Worsening of Fbrosis by Histology (Evaluated by BICR) After 52 Weeks
Description: Participants with ≥2 point improvement in the NAS with ≥1 point improvement in inflammation or ballooning without worsening of fibrosis were assessed with the NASH CRN scoring system (evaluated by BICR). The NAS was calculated as the unweighted sum of the scores and ranges from 0-8 (highest activity).
Time Frame: Week 52
Population: as for outcome 4
Measure: Number; unit: Percentage of Participants
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
Number analyzed (Participants) | 18 | 21 | 17 | 17
Percentage of Participants | 33.3 | 47.6 | 35.3 | 29.4
Statistical Analysis 1: Comparison: MK-3655 50 mg vs Placebo; Test type: Other; p = 0.9174, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 1.6, 95% CI 2-sided [-28.6 to 32.6] — Difference=% 50 mg minus % Placebo
Statistical Analysis 2: Comparison: MK-3655 100 mg vs Placebo; Test type: Other; p = 0.2720, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 18.5, 95% CI 2-sided [-14.5 to 47.1] — Difference=% 100 mg minus % Placebo
Statistical Analysis 3: Comparison: MK-3655 300 mg vs Placebo; Test type: Other; p = 0.7586, Miettinen and Nurminen's method; [statistical method as in outcome 1, analysis 1]; Difference in Percentages = 5.3, 95% CI 2-sided [-26.7 to 37.3] — Difference= % 300 mg minus % Placebo

ADVERSE EVENTS:
Time Frame: Up to 64 weeks
Description: All-cause mortality population included all enrolled participants. Serious Adverse Events (SAEs) and non-serious AEs population included all participants who received at least 1 dose of study drug.
Arm/Group | MK-3655 50 mg | MK-3655 100 mg | MK-3655 300 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/48 | 0/46 | 0/44
Serious Adverse Events (participants affected / at risk) | 1/45 | 1/47 | 1/46 | 8/44
Other Adverse Events (participants affected / at risk) | 19/45 | 26/47 | 27/46 | 21/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3655 50 mg (N=45) | MK-3655 100 mg (N=47) | MK-3655 300 mg (N=46) | Placebo (N=44)
Sinoatrial block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-3655 50 mg (N=45) | MK-3655 100 mg (N=47) | MK-3655 300 mg (N=46) | Placebo (N=44)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 7 (7) | 5 (5) | 3 (5)
Nausea (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (2) | 4 (4)
Pyrexia (General disorders) | 2 (4) | 2 (2) | 2 (2) | 4 (5)
COVID-19 (Infections and infestations) | 4 (4) | 9 (11) | 5 (6) | 5 (5)
Influenza (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 2 (2) | 4 (6) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (3) | 2 (2) | 1 (1) | 1 (1)
Weight increased (Investigations) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 5 (5) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 7 (11) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2) | 3 (3) | 4 (6) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 3 (4)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 5 (6) | 3 (4)
Hypertension (Vascular disorders) | 2 (2) | 6 (8) | 6 (7) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity was not directed by the Sponsor, the investigator agreed to submit all manuscripts or abstracts to the Sponsor before submission. This allowed the Sponsor to protect proprietary information and to provide comments.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-24): https://cdn.clinicaltrials.gov/large-docs/23/NCT04583423/Prot_SAP_000.pdf